CLINICAL TRIAL: NCT05141370
Title: Assessment of a Hand-held Femtosecond Laser to Perform Anterior Capsulorhexis During Cataract Surgery
Brief Title: Assessment of a Femtosecond Laser to Perform Capsulorhexis During Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilasis Laser (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A02331-40
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cataract Surgery
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hand-held femtosecond laser (Experimental): Anterior capsulorhexis will be performed with a hand-held femtosecond laser named CATSYS.
  Interventions: Device: cataract surgery with CATSYS

INTERVENTIONS:
Device: cataract surgery with CATSYS — patient diagnosed with cataract requiring surgery will have an anterior capsulorhexis with CATSYS

SUMMARY:
This study is a Pre-market first-in-man clinical investigation to validate performance of a hand-held femtosecond laser named CATSYS.

DETAILED DESCRIPTION:
Interventional, prospective, longitudinal (follow-up: 30 ± 10 days), single-arm, single center, open trial. The "first-in-man" character of this investigation relies on the ergonomics of CATSYS (handpiece), and not on the laser technique, which is similar to other FLACS.

The purpose of the clinical investigation is to document the compliance of the investigational medical device with the general requirements of performance, safety and clinical benefit, in order to complete existing data and obtaining CE-mark for CATSYS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cataract requiring surgery according to current guidelines;
* Eligible to lens removal by phacoemulsification and replacement by a prosthetic lens under local anesthesia;
* Who have been informed and gave informed consent to participate in the study.

Exclusion Criteria:

* Eye with an anterior chamber depth < 2.5 mm or > 3.8 mm;
* Corneal disease or pathology that precludes applanation of the cornea or transmission of laser wavelength or distortion of laser light;
* Eye with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally;
* Patient with residual, recurrent, active ocular or eyelid disease, including any corneal abnormality (for example, recurrent corneal erosion, severe basement membrane disease) in either eye;
* History of steroid-responsive rise in IOP, glaucoma, or preoperative IOP>21 mm Hg in either eye;
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, pseudoexfoliation syndrome, etc;
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye;
* Any recent penetrating incision of the eyeball;
* Tilt of lens > 7;
* Presence of any obstacle that may interfere with the stabilization of the device on the limbus: pterygium, limbic tumor, etc;
* Pregnant or lactating woman;
* Patient with any contra-indication to neosynephrine, tropicamide and oxybuprocaïne;
* Patient presenting any contraindications to cataract surgery under local anesthesia (ex: allergy to anesthetic drops; neurodegenerative disease; schizophrenia; severe anxiety; etc.);
* Patient who participates to another clinical trial (except observational studies), or in the exclusion period of another clinical trial;
* Patient under guardianship, trusteeship or deprived of liberty;
* Patient not affiliated to the French social security system;
* Patient unable to participate in the study for psychiatric, cognitive or linguistic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Continuity of the capsulorhexis (success / failure) | During surgery
  Success achieved if:
  * the anterior capsule is completely cut (rhexis is free floating or easy to remove)
  * AND there are no peripheric tears that can generate the rupture of the capsule at the end of rhexis removal.

SECONDARY OUTCOMES:
Adverse device effects | 3 to 5 days after surgery
  Collection of adverse device effects by the investigator on the retina, on the cornea, on the posterior capsula and other adverse device events
Adverse events | 3 to 5 days post-surgery;
  Collection by the investigator of other adverse events
Ocular adverse events | 30 ± 10 days post-surgery.
  Collection by the investigator of ocular adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Opthalmologique Sourdille Atlantique, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No